CLINICAL TRIAL: NCT01875289
Title: Efficacy of a Modified Obturator Nerve Block Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Andreas Sandner-Kiesling , MD, Prof. Dr. med. univ., Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VOB-Studie EK 25-387 ex 12/13
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Hip Surgery; Knee Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ropivacain (Experimental): Local anaesthesia
  Interventions: Procedure: obturator nerve block
- NaCl 0.9% (Placebo Comparator): Saline
  Interventions: Procedure: obturator nerve block

INTERVENTIONS:
Procedure: obturator nerve block

SUMMARY:
Efficacy of a modified obturator nerve block technique by using only a single morphological landmark, a double-blinded randomised pilot study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists 1-3, older than 18 y, cooperative patient

Exclusion Criteria:

* infection, neuromuscular deficits of the lower extremities,pregnancy, neurologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Adductor strengths | pre operative, 30 minutes before start surgery
  Adductor muscle strength is measured with a sphygmomanometer. Patients are instructed to squeeze a blod pressure cuff, already inflated to 40 mm Hg, between their extended knees. The maximal sustained pressure is taken as the baseline adductor strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Austria

REFERENCES:
- [Background] Feigl GC, Ulz H, Pixner T, Dolcet C, Likar R, Sandner-Kiesling A. Anatomical investigation of a new vertical obturator nerve block technique. Ann Anat. 2013 Jan;195(1):82-7. doi: 10.1016/j.aanat.2012.05.008. Epub 2012 Aug 10. PMID 22951254